CLINICAL TRIAL: NCT01754922
Title: Effects of Deployment Exposures on Cardiopulmonary and Autonomic Function
Acronym: AirHzds
Status: Completed | Type: Observational
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: F1079-P; 1I21RX001079-01A (Other Grant/Funding Number: VA ORD RR&D); 1I21RX001079-01 (NIH)
Record Dates: First submitted 2012-12-18; First posted 2012-12-21 (Estimated); Results first posted 2016-10-26 (Estimated); Last update posted 2017-02-28 (Actual); Status verified 2017-01

CONDITIONS: Abnormality, Respiratory System; Autonomic Nervous System
Keywords: exercise tolerance; Veterans; operation enduring freedom; operation Iraqi freedom
MeSH Terms: conditions — Respiratory System Abnormalities

STUDY DESIGN:
Time Perspective: Cross-Sectional
Biospecimen Retention: None Retained — No biospecimens will be collected
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Exposed: Veterans deployed to OEF/OIF/OND and environmentally exposed to high levels of particulate matter
- Control: OEF/OIF/OND Veterans deployed to regions other than Southwest Asia

SUMMARY:
Following deployment to Operations Enduring and Iraqi Freedom and Operation New Dawn (OEF/OIF/OND), Veterans report breathing problems, difficulty exercising and other symptoms. These symptoms may be related to deployment exposures, such as regional dust and sand, smoke from burning trash, and local industry. Studies have reported poor air quality, but very little is known about the effect that exposure to this polluted air may have on Veterans' short- and long-term health. Investigators will determine whether deployment-related exposures have affected respiratory and nervous system function in these Veterans - data that may then be used to guide rehabilitation. Ultimately, the investigators' long-term goal is to prevent the development of chronic respiratory conditions in this group of OEF/OIF/OND Veterans.

DETAILED DESCRIPTION:
Evidence is clear that Veterans deployed to Operations Enduring and Iraqi Freedom and Operation New Dawn (OEF/OIF/OND) have been exposed to high levels of particulate matter (PM) that exceeded environmental, occupational and military exposure guidelines. PM exposure is acknowledged as a risk factor for cardiovascular morbidity and mortality, and can increase the risk of and exacerbate airway disease. The reviewed epidemiology indicates a high prevalence of newly reported respiratory symptoms in OEF/OIF/OND Veterans that has significantly affected their deployment duties, including their physical exertion capability. Despite these retrospective data and limited air sampling reports, prospective studies are lacking. This pilot study will evaluate cardiorespiratory and autonomic function in OEF/OIF/OND Veterans as compared to Veterans never deployed to the region.

To evaluate cardiopulmonary function, each Veteran will undergo a standardized exercise challenge and bronchodilator spirometry. To evaluate autonomic nervous system function, investigators will examine indices of heart rate variability and cardiovascular reflex regulation (e.g. baroreflex sensitivity and cerebral autoregulation) during a variety of tasks.

Data derived from this pilot project will yield important insight on the extent and severity of cardiorespiratory and/or autonomic impairments - data that may provide intervention points for attenuating long-term adverse outcomes such as pulmonary and cardiovascular disease. Through early identification, treatment options (e.g. exercise therapy, pharmaceutical) may be implemented to enhance physiological function, with the goal of helping to alleviate symptoms and reduce chronic disease risk.

ELIGIBILITY:
Inclusion Criteria:

* Male and female Veterans between 18 - 55 years of age will be identified and screened for this study.
* Two study cohorts will be recruited and attempts will be made to match group composition on age, body mass index and smoking history.
* Veterans assigned to the Exposed group must have been deployed to OEF/OIF for a minimum of 90 consecutive days.
* The Control group will consist of Veterans never deployed to Southwest Asia (i.e. OEF/OIF, Persian Gulf War) but were deployed during the same time period.
* Each Veteran will complete a detailed exposure history questionnaire to confirm and support their group assignment.

Exclusion Criteria:

Participants must not meet any of the contraindications to exercise testing as described in the joint statement from the American College of Cardiology and American Heart Association. Also, individuals with history of any of the following will also be excluded:

* asthma (pre-military)
* cardiovascular disease
* neurological impairment/disorder
* pregnant
* uncontrollable hypertension (SBP > 160; DBP > 100)
* or have suffered severe/moderate traumatic brain injury within the last three years
* eye/chest/abdominal surgery in last 3 months
* tuberculosis exposure to self or household member
* history of aneurysm or collapsed lung
* history of detached retina
* stroke or heart attack in the last 3 months
* and history of coughing up blood in last three months

(With the exception of hypertension and pregnancy (urine test), all exclusion criteria will be determined via self-report)

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Community sample, outpatient clinic
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2013-11; Primary Completion 2015-08 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Joseph Falvo, PhD, Principal Investigator — East Orange Campus of the VA New Jersey Health Care System, East Orange, NJ
Locations (1):
- East Orange Campus of the VA New Jersey Health Care System, East Orange, NJ, East Orange, New Jersey, United States

REFERENCES:
- See also: PI contact information and study site information — http://www.warrelatedillness.va.gov/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Exposed | Control
Started | 32 | 18
Completed | 32 | 17
Not Completed | 0 | 1
Not completed — Adverse Event | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Control: Veterans deployed to regions other than Iraq or Afghanistan or non-deployed
- Total: Total of all reporting groups
Arm/Group | Exposed | Control | Total
Number analyzed (Participants) | 32 | 18 | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.8 (8.1) | 33.2 (9.7) | 34.6 (8.7)
Gender [Count of Participants; unit: Participants]
  Female | 6 | 5 | 11
  Male | 26 | 13 | 39
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 7 | 14 | 21
  White | 23 | 4 | 27
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 32 | 18 | 50
Tobacco Pack Years [Mean (Standard Deviation); unit: Pack Years] | 1.45 (3.42) | 1.65 (5.2) | 1.5 (4.08)

OUTCOME MEASURES:

1. Primary Outcome: FEV1
Description: Forced expiratory volume in 1 second (FEV1) measured before and after an exercise challenge
Time Frame: Pre/post exercise; cross-sectional
Measure: Mean (Standard Deviation); unit: percentage of predicted normal values
Groups:
- Control: Veterans deployed to regions other than Iraq and Afghanistan or non-deployed
Arm/Group | Exposed | Control
Number analyzed (Participants) | 32 | 18
percentage of predicted normal values
  Pre-Exercise FEV1 | 0.94 (.16) | 1.08 (.16)
  Post-Exercise FEV1 | 0.95 (0.18) | 1.09 (0.17)

2. Primary Outcome: VO2 Peak
Description: Maximal oxygen consumption measured during exercise
Time Frame: At peak exercise; cross-sectional
Population: 4 participants were excluded due to failure to meet maximal exercise criteria (3 from exposed, 1 from control). Therefore, we removed these individuals from the final analysis.
Measure: Mean (Standard Deviation); unit: ml/min/kg
Arm/Group | Exposed | Control
Number analyzed (Participants) | 29 | 17
ml/min/kg | 33.79 (8.6) | 34.49 (10.4)

3. Primary Outcome: Heart Rate Variability
Description: Ratio of low-frequency to high-frequency power for heart rate variability
Time Frame: Resting baseline; cross-sectional
Population: Signal quality of the the electrocardiogram was poor for 3 individuals; therefore, their data were removed from final analysis.
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Exposed | Control
Number analyzed (Participants) | 29 | 18
Ratio | 2.02 (1.7) | 1.13 (1.1)

ADVERSE EVENTS:
Groups:
- Control: OEF/OIF/OND Veterans deployed to regions other than Southwest Asia or non-deployed
Arm/Group | Exposed | Control
Serious Adverse Events (participants affected / at risk) | 0/32 | 1/18
Other Adverse Events (participants affected / at risk) | 0/32 | 0/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Exposed (N=32) | Control (N=18)
Psychiatric emergency (Psychiatric disorders) | 0 (0) | 1 (1) — Participant experienced a psychiatric emergency upon arrival for a laboratory visits. A staff psychologist evaluated the participant and admitted to the emergency room for further clinical care.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes